CLINICAL TRIAL: NCT07089849
Title: HIV Testing in Community Health Center Dental Clinics
Acronym: TEETH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-43301; 5UH3DE031249-04 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: HIV
Keywords: Rapid HIV test; Referral for HIV test; Community Health Center Dental Clinics; Behavioral Model for Vulnerable Populations
MeSH Terms: interventions — Referral and Consultation; HIV Testing

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial among dental clinics (n=4)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid HIV Testing (Experimental): Dental clinics randomized into this arm will offer Rapid HIV Testing at the patient's dental visit.
  Interventions: Other: Rapid HIV testing
- Referral HIV Testing (Active Comparator): Dental clinics randomized into this arm will offer a referral for HIV Testing during the patient's dental visit.
  Interventions: Other: Referral for HIV testing

INTERVENTIONS:
Other: Rapid HIV testing — At the designated sites for RHT, providers will offer RHT to patients as part of their dental routine care.
  Arms: Rapid HIV Testing
Other: Referral for HIV testing — At the designated sites for HIV testing referral, providers will offer an HIV test referral to the affiliated CHC laboratory to patients as part of their dental routine care.
  Arms: Referral HIV Testing

SUMMARY:
This is a cluster randomized trial among dental clinics (n=4) to evaluate whether rapid HIV testing (RHT) during dental visits improves HIV testing rates compared to referral for laboratory HIV testing. Clinics will be randomized to either RHT or referral for HIV testing for a nine-month period - HIV testing will be offered to n~6700 patients by ~ 15 dental providers (dentists and dental hygienists). Outcomes will be assessed using electronic health record reports (EHR), which will include the completion rates of HIV testing among dental patients (84 days after dental visit) and the frequency at which dental providers offer HIV testing (Upon completion of the 9-month testing period).

The objectives of this study are to:

* Compare the effectiveness of on-site rapid HIV testing versus referral to a CHC lab in increasing HIV test completion within 84 days of a dental clinic visit, using EHR data.
* Assess the sustainability of the HIV testing protocol by evaluating changes in dental clinic HIV testing rates over time.

ELIGIBILITY:
Inclusion Criteria:

Community health center:

* Must be located in Suffolk County in Massachusetts.
* Must provide dental care services.
* Must possess the infrastructure necessary for laboratory-based HIV testing and counseling or have an affiliation with a laboratory that provides these service.

Provider:

* Dental care provider working at a participating community health center during the study period.

Patient:

* Be 18 years of age or older.
* Receive dental care at a participating community health center during the study period.

Exclusion Criteria:

Patient:

* Self-report to be HIV positive at the time of the RHT/ referral.
* Had an HIV test within 12 months (self-report or documented in EHR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6715 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
HIV Test Completed | 84 days
  The number of dental patients completing at least one HIV test within 84 days of their dental visit abstracted from the Electronic Health Records (EHR).
Sustainability | 9 months
  The number of dental patients completing at least one HIV test within 9 months of their dental visit abstracted from the Electronic Health Records (EHR).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Henshaw, DDS MPH, Principal Investigator — Boston University Goldman School of Dental Medicine; Curt Beckwith, MD FACP FIDSA, Principal Investigator — The Miriam Hospital/Rhode Island Hospital
Locations (4):
- United States (4):
  - South End Community Health Center, Boston, Massachusetts
  - Uphams Corner Health Center, Boston, Massachusetts
  - East Boston Neighborhood Health, Boston, Massachusetts
  - Geiger Gibson Community Health Center, Dorchester, Massachusetts

IPD SHARING:
Plan to Share IPD: No